CLINICAL TRIAL: NCT01554176
Title: A Phase IIa, Multicenter, Randomized, Placebo-Controlled Clinical Trial to Evaluate the Safety and Efficacy of MK-6096 for Treatment Augmentation in Patients With Major Depressive Disorder
Brief Title: Safety and Efficacy of MK-6096 as Adjunctive Therapy in Participants With Major Depressive Disorder And Partial Response to Antidepressant Monotherapy (MK-6096-022)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6096-022; 2011-005200-15 (EudraCT Number)
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Major Depressive Disorder, Recurrent
Keywords: Current depressive episode; moderate to severe
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence | interventions — MK-6096

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Filorexant 10 mg (Treatment Phase) (Experimental): Treatment Phase: Participants in this group were administered filorexant 10 mg once daily at bedtime for 6 weeks.
  Interventions: Drug: Filorexant
- Placebo (Treatment Phase) (Placebo Comparator): Treatment Phase: Participants in this group were administered placebo once daily at bedtime for 6 weeks.
  Interventions: Drug: Placebo
- Filorexant 10 mg/Filorexant 10 mg (Run-out Phase) (Experimental): Run-out Phase: Following completion of the 6-week treatment phase, participants in this group were administered filorexant 10 mg once daily at bedtime for 2 weeks. Participants in this group had received filorexant 10 mg once daily during the treatment phase.
  Interventions: Drug: Filorexant
- Filorexant 10 mg/Placebo (Run-out Phase) (Placebo Comparator): Run-out Phase: Following completion of the 6-week treatment phase, participants in this group were administered placebo once daily at bedtime for 2 weeks. Participants in this group had received filorexant 10 mg once daily during the treatment phase.
  Interventions: Drug: Filorexant; Drug: Placebo
- Placebo/Placebo (Run-out Phase) (Placebo Comparator): Run-out Phase: Following completion of the 6-week Treatment Phase, participants in this group were administered placebo once daily at bedtime for 2 weeks. Participants in this group had received placebo once daily during the Treatment Phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Filorexant — Filorexant, one 10 mg tablet, orally, once daily at bedtime
  Other Names: MK-6096
  Arms: Filorexant 10 mg (Treatment Phase); Filorexant 10 mg/Filorexant 10 mg (Run-out Phase); Filorexant 10 mg/Placebo (Run-out Phase)
Drug: Placebo — Placebo, one tablet, orally, once daily at bedtime
  Arms: Filorexant 10 mg/Placebo (Run-out Phase); Placebo (Treatment Phase); Placebo/Placebo (Run-out Phase)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of filorexant (MK-6096) versus placebo as adjunctive treatment for major depressive disorder (MDD), in participants who are partial responders to antidepressant monotherapy with one of identified selective serotonin reuptake inhibitors (SSRIs) or serotonin norepinephrine reuptake inhibitors (SNRIs), or bupropion. The primary hypothesis of the study is that filorexant is superior to placebo as augmentation therapy with respect to change from baseline to Week 6 in the Montgomery Asberg Depression Rating Scale (MADRS) total score.

DETAILED DESCRIPTION:
Participants will continue to take their pretrial antidepressant medication as prescribed throughout the trial. Participants will be randomized in a 1:1 ratio to receive filorexant or placebo for a 6-week treatment period. Following completion of the treatment period, participants will enter a 2-week double-blind run-out period. During the run-out period, participants who received placebo in the 6-week treatment period will continue to receive placebo and participants who received filorexant in the 6-week treatment period will be randomized to receive either filorexant or placebo in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Participant is (a) male or (b) female and not of reproductive potential, or (c) female of reproductive potential has a serum beta-hCG level consistent with the nongravid state at screening and agrees to use acceptable contraception;
* Current primary diagnosis of recurrent major depressive disorder, without psychotic features, with a current moderate or severe depressive episode;
* Duration of the current major depressive episode must be at least 2 months but no more than 18 months at Screening;
* Participant has undergone an adequate trial of an antidepressant (one of identified SSRIs or SNRIs, or bupropion) for the current depressive episode.

Key Exclusion Criteria:

* Current primary psychiatric diagnosis other than major depression;
* Lifetime diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder, or other psychotic disorder;
* Alcohol or other substance abuse or dependence (excluding nicotine);
* Clinically significant abnormality or disease of the central nervous system (including dementia and other cognitive disorders or traumatic brain injury);
* Imminent risk of self-harm or of harm to others;
* Participant is a psychiatric inpatient;
* Participant has been on continuous antidepressant treatment for >18 months prior to Screening visit;
* Inadequate response to more than 3 adequate antidepressant trials (including the current antidepressant treatment trial) for treatment of the current depressive episode;
* Participant ever received electroconvulsive therapy, transcranial magnetic stimulation, or vagal nerve stimulation for treatment of depression;
* History of narcolepsy, cataplexy, circadian rhythm disorder, parasomnia, sleep-related breathing disorder, restless legs syndrome, periodic limb movement disorder, excessive daytime sleepiness or difficulty sleeping due to a medical condition;
* Clinical, laboratory, or electrocardiogram (ECG) evidence of significant systemic disease;
* Cardiovascular event (e.g., myocardial infarction) or procedure (e.g., coronary artery bypass surgery) within 3 months of study;
* History of malignancy ≤5 years prior to study, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer;
* Body Mass Index >40 kg/m^2;
* Pregnancy, breast-feeding, or expecting to become pregnant.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2012-05-18 (Actual); Primary Completion 2013-09-03 (Actual); Study Completion 2013-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Connor KM, Ceesay P, Hutzelmann J, Snavely D, Krystal AD, Trivedi MH, Thase M, Lines C, Herring WJ, Michelson D. Phase II Proof-of-Concept Trial of the Orexin Receptor Antagonist Filorexant (MK-6096) in Patients with Major Depressive Disorder. Int J Neuropsychopharmacol. 2017 Aug 1;20(8):613-618. doi: 10.1093/ijnp/pyx033. PMID 28582570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant in the Filorexant 10 mg (Treatment Phase) arm did not receive study drug and was discontinued from the study; the reason given for discontinuation is given as "non-compliance with study drug".
Pre-assignment Details: During the 1-2 week screening period participants will be evaluated to determine if they meet study entry criteria. The screening period will serve as a wash-out period for participants taking prohibited medications.
Period: Treatment Phase
Arm/Group | Filorexant 10 mg (Treatment Phase) | Placebo (Treatment Phase) | Filorexant 10 mg/Filorexant 10 mg (Run-out Phase) | Filorexant 10 mg/Placebo (Run-out Phase) | Placebo/Placebo (Run-out Phase)
Started | 65 | 64 | 0 | 0 | 0
Treated | 64 | 64 | 0 | 0 | 0
Completed | 57 | 59 | 0 | 0 | 0
Not Completed | 8 | 5 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0
Not completed — Adverse event, non-fatal | 1 | 1 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0 | 0
Period: Run-out Phase
Arm/Group | Filorexant 10 mg (Treatment Phase) | Placebo (Treatment Phase) | Filorexant 10 mg/Filorexant 10 mg (Run-out Phase) | Filorexant 10 mg/Placebo (Run-out Phase) | Placebo/Placebo (Run-out Phase)
Started | 0 | 0 | 29 | 28 | 59
Treated | 0 | 0 | 29 | 28 | 59
Completed | 0 | 0 | 29 | 27 | 59
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Filorexant 10 mg (Treatment Phase) | Placebo (Treatment Phase) | Total
Number analyzed (Participants) | 65 | 64 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.8 (12.4) | 50.0 (10.3) | 48.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a 10-item clinician-rated instrument for evaluating severity of symptoms of depression. Each item is rated on a scale from 0 to 6, with total scores ranging from 0 to 60; higher scores correspond to greater symptom severity. The reported measure is the mean change from baseline to Week 6 of the Treatment Phase; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Week 6
Population: Full Analysis Set (FAS) - population included participants who took ≥1 dose of study drug and had a baseline and Week 6 value.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filorexant 10 mg (Treatment Phase) | Placebo (Treatment Phase)
Number analyzed (Participants) | 58 | 61
score on a scale
  Baseline | 30.3 (4.6) | 31 (4.3)
  Change at Week 6 | -11 (9.5) | -10.3 (8.2)
Statistical Analysis 1: Comparison: Filorexant 10 mg (Treatment Phase) vs Placebo (Treatment Phase); Number of participants included for calculation of mean ± SD baseline and mean ± SD change from baseline MADRS Total Score is 119. Constrained longitudinal data analysis (cLDA) model uses efficacy Full Analysis Set (FAS) population (number of participants: filorexant 10 mg - 64, placebo - 64; total number of participants in cLDA analysis - 128); Test type: Superiority or Other; p = 0.679, cLDA — cLDA model included terms for treatment, time, the interaction of time by treatment, severity of disease (Hamilton Depression Rating Scale, 17-items [HAM-D17] ≤20, >20) and insomnia severity index (ISI ≤14, >14); Difference in least squares means = -0.7, 95% CI 2-sided [-3.8 to 2.5]

2. Secondary Outcome: Change From Baseline to Week 6 in MADRS Total Score Excluding the Sleep Item
Description: The MADRS is a 10-item clinician-rated instrument for evaluating severity of symptoms of depression. Each item is rated on a scale from 0 to 6, with higher scores indicating greater symptom severity. The total score ranged from 0 to 54, with higher scores corresponding to greater symptom severity. This measure considered 9 of the 10 MADRS items: apparent sadness, reported sadness, inner tension, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. It excluded "reduced sleep." The reported measure is the mean change from baseline to Week 6 of the Treatment Phase; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Week 6
Population: Full Analysis Set (FAS) - population included participants who took ≥1 dose of study drug and had a baseline and Week 6 MADRS score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filorexant 10 mg (Treatment Phase) | Placebo (Treatment Phase)
Number analyzed (Participants) | 58 | 61
score on a scale
  Baseline | 26.5 (4.1) | 27.2 (4.1)
  Change at Week 6 | -9.5 (8.5) | -9.1 (7.4)
Statistical Analysis 1: Comparison: Filorexant 10 mg (Treatment Phase) vs Placebo (Treatment Phase); Pairwise Comparison: Filorexant 10 mg vs. Placebo; Test type: Superiority or Other; p = 0.820, cLDA — [p-value comment as in outcome 1, analysis 1]; Difference in least squares means = -0.3, 95% CI 2-sided [-3.2 to 2.5]

3. Secondary Outcome: Change From Baseline to Week 6 in the Hamilton Depression Rating Scale, 17-item Version (HAM-D17) Bech Subscale Score
Description: The HAM-D, an instrument for evaluating severity of symptoms of depression, was completed by the participant. The instrument used in this study was the 17-item version (HAM-D17). The Bech subscale of the HAM-D17 is composed of 6 identified items out of the 17 items rated. Each item is rated on either a 3-point scale (0 to 2) or a 5-point scale (0 to 4). Total score ranged from 0 to 22, with a higher score indicating greater symptom severity. The following symptoms were rated on a 5-point scale (0-4): depressed mood, low self-esteem (guilt), work and interests, psychomotor retardation, and anxiety (psychic). The following symptom was rated on a 3-point scale (0-2): somatic symptoms (general). The reported measure is the change from baseline to Week 6 of the Treatment Phase; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Week 6
Population: Full Analysis Set (FAS) - population included participants who took ≥1 dose of study drug and had a baseline and Week 6 HAM-D17 Beck Subscale score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filorexant 10 mg (Treatment Phase) | Placebo (Treatment Phase)
Number analyzed (Participants) | 56 | 61
score on a scale
  Baseline | 13.1 (2.4) | 13.0 (2.1)
  Change at Week 6 | -4.7 (4.8) | -4.2 (4.0)
Statistical Analysis 1: Comparison: Filorexant 10 mg (Treatment Phase) vs Placebo (Treatment Phase); Pairwise Comparison: Filorexant 10 mg vs. Placebo; Test type: Superiority or Other; p = 0.701, cLDA — [p-value comment as in outcome 1, analysis 1]; Difference in least squares means = -0.3, 95% CI 2-sided [-1.9 to 1.3]

4. Secondary Outcome: Percentage of Participants With HAM-D17 Remission (HAM-D17 Total Score ≤7) at Week 6
Description: The HAM-D, an instrument for evaluating severity of symptoms of depression, was completed by the participant. The instrument used in this study was the 17-item version (HAM-D17). Each item is rated on either a 3-point scale (0 to 2) or a 5-point scale (0 to 4), with higher scores indicating greater symptom severity. Total score ranged from 0 to 54. The following symptoms were rated on a 5-point scale (0-4): depressed mood, low self-esteem (guilt), suicidal thoughts, work and interests, psychomotor retardation, psychomotor agitation, anxiety (psychic), anxiety (somatic), and hypochondriasis (somatization). The following symptoms were rated on a 3-point scale (0-2): insomnia (initial), insomnia (middle), insomnia (late), gastrointestinal symptoms (appetite), somatic symptoms (general), sexual disturbances, insight, and weight loss. A participant with HAM-D17 total score ≤7 at Week 6 of the Treatment Phase was defined to have achieved HAM-D17 remission.
Time Frame: Week 6
Population: Full Analysis Set (FAS) - population included participants who took ≥1 dose of study drug and had a baseline and Week 6 HAM-D17 score.
Measure: Number; unit: percentage of participants
Arm/Group | Filorexant 10 mg (Treatment Phase) | Placebo (Treatment Phase)
Number analyzed (Participants) | 56 | 61
percentage of participants | 21.4 | 9.8
Statistical Analysis 1: Comparison: Filorexant 10 mg (Treatment Phase) vs Placebo (Treatment Phase); Pairwise Comparison: Filorexant 10 mg vs. Placebo; Test type: Superiority or Other; p = 0.0965, Generalized Linear Mixed Effects Model — Generalized linear mixed effects model included terms for treatment, time, treatment-by-time interaction; Estimated Odds Ratio = 2.5, 95% CI 2-sided [0.8 to 7.3]

5. Primary Outcome: Number of Participants With an Adverse Event (AE) During Treatment Phase
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with study drug administration, is also an AE. Participants with one or more AEs during the treatment phase (up to study Week 6) are counted once in this summary.
Time Frame: Up to Week 6
Population: All Participants as Treated (APaT): Population includes participants who took ≥1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Filorexant 10 mg (Treatment Phase) | Placebo (Treatment Phase)
Number analyzed (Participants) | 64 | 64
Participants | 27 | 17
Statistical Analysis 1: Comparison: Filorexant 10 mg (Treatment Phase) vs Placebo (Treatment Phase); Estimated parameter is between-group difference in percentage of participants with an AE = percentage (filorexant 10 mg) - percentage (placebo) for participants with one or more AE; Test type: Superiority or Other; Between-group comparison of AE incident rate; Difference in percentage incidence = 15.6, 95% CI 2-sided [-0.9 to 31.4]

6. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE During Treatment Phase
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with study drug administration, is also an AE. Participants who discontinued study drug treatment due to an AE during the treatment phase (up to study Week 6) are counted once in this summary.
Time Frame: Up to Week 6
Population: All Participants as Treated (APaT): Population includes participants who took ≥1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Filorexant 10 mg (Treatment Phase) | Placebo (Treatment Phase)
Number analyzed (Participants) | 64 | 64
Participants | 1 | 1
Statistical Analysis 1: Comparison: Filorexant 10 mg (Treatment Phase) vs Placebo (Treatment Phase); Estimated parameter is between-group difference in percentage of participants discontinued from study drug due to an AE = percentage (filorexant 10 mg) - percentage (placebo); Test type: Superiority or Other; Between-group comparison of incidence rate of drug discontinuation due to AE; Difference in percentage incidence = 0, 95% CI 2-sided [-7 to 7]

7. Primary Outcome: Number of Participants With an AE During Run-out Phase
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with study drug administration, is also an AE. Participants with one or more AEs during the 2-week run-out phase and/or during the 2-week follow up after the last dose of study drug, are counted once in this summary.
Time Frame: From first run-out dose (following Week 6 visit) up to 14 days after last dose of study drug (approximately 4 weeks)
Population: All Participants as Treated (APaT): Population includes participants who took ≥1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Filorexant 10 mg/Filorexant 10 mg (Run-out Phase) | Filorexant 10 mg/Placebo (Run-out Phase) | Placebo/Placebo (Run-out Phase)
Number analyzed (Participants) | 29 | 28 | 59
Participants | 6 | 3 | 9

8. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE During Run-out Phase
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) or a preexisting condition which is temporally associated with study drug administration, is also an AE. Participants who discontinued study drug treatment due to an AE during the 2-week run-out phase are counted once in this summary.
Time Frame: From first run-out dose (following Week 6 visit) up to Week 8 (2 weeks)
Population: All Participants as Treated (APaT): Population includes participants who took ≥1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Filorexant 10 mg/Filorexant 10 mg (Run-out Phase) | Filorexant 10 mg/Placebo (Run-out Phase) | Placebo/Placebo (Run-out Phase)
Number analyzed (Participants) | 29 | 28 | 59
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment Phase: Up to Week 6 Run-out Phase: From first run-out dose (following Week 6 visit) up to 14 days after last dose of study drug (approximately 4 weeks)
Description: All Participants as Treated (APaT): Population includes participants who took ≥1 dose of study drug.
Arm/Group | Filorexant 10 mg (Treatment Phase) | Placebo (Treatment Phase) | Filorexant 10 mg/Filorexant 10 mg (Run-out Phase) | Filorexant 10 mg/Placebo (Run-out Phase) | Placebo/Placebo (Run-out Phase)
Serious Adverse Events (participants affected / at risk) | 1/64 | 0/64 | 0/29 | 0/28 | 1/59
Other Adverse Events (participants affected / at risk) | 13/64 | 7/64 | 3/29 | 1/28 | 1/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Filorexant 10 mg (Treatment Phase) (N=64) | Placebo (Treatment Phase) (N=64) | Filorexant 10 mg/Filorexant 10 mg (Run-out Phase) (N=29) | Filorexant 10 mg/Placebo (Run-out Phase) (N=28) | Placebo/Placebo (Run-out Phase) (N=59)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Filorexant 10 mg (Treatment Phase) (N=64) | Placebo (Treatment Phase) (N=64) | Filorexant 10 mg/Filorexant 10 mg (Run-out Phase) (N=29) | Filorexant 10 mg/Placebo (Run-out Phase) (N=28) | Placebo/Placebo (Run-out Phase) (N=59)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 5 (5) | 1 (1) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.